CLINICAL TRIAL: NCT04754022
Title: An International, Multi-centre, Randomized Controlled Trial to Assess Transfusion Thresholds in Younger Patients Undergoing Cardiac Surgery
Brief Title: Transfusion Requirements in Younger Patients Undergoing Cardiac Surgery
Acronym: TRICS-IV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRICS-IV
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Disorder; Heart; Postoperative; Cardiac Surgery
Keywords: Cardiac Surgery; Transfusion
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restrictive Transfusion Strategy (Active Comparator): Patients will receive a RBC transfusion if their Hb concentration is <75 g/L (<7.5 g/dL; <4.7mmol/L) intraoperatively and/or postoperatively.
  Interventions: Other: Restrictive Transfusion Strategy
- Liberal Transfusion Strategy (Active Comparator): Patients will receive a RBC transfusion if their Hb concentration is <95 g/L (<9.5 g/dL; <5.9mmol/L) intraoperatively, or postoperatively in the ICU; and/or <85 g/L (< 8.5 g/dL; <5.3mmol/L) on the ward.
  Interventions: Other: Liberal transfusion strategy

INTERVENTIONS:
Other: Restrictive Transfusion Strategy — Patients will receive a RBC transfusion if their Hb concentration is <75 g/L (<7.5 g/dL; <4.7mmol/L) intraoperatively and/or postoperatively.
  Arms: Restrictive Transfusion Strategy
Other: Liberal transfusion strategy — Patients will receive a RBC transfusion if their Hb concentration is <95 g/L (<9.5 g/dL; <5.9mmol/L) intraoperatively, or postoperatively in the ICU; and/or <85 g/L (< 8.5 g/dL; <5.3mmol/L) on the ward.
  Arms: Liberal Transfusion Strategy

SUMMARY:
TRICS-IV is an international, multi-centre, open-label randomized controlled trial of two commonly used transfusion strategies in moderate to high risk patients who are 65 years of age or younger undergoing cardiac surgery on cardiopulmonary bypass, using a superiority trial design.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤65 years of age
2. Planned cardiac surgery using cardiopulmonary bypass
3. Informed consent obtained
4. Preoperative European System for Cardiac Operative Risk Evaluation (EuroSCORE I) of 6 or more

Exclusion Criteria:

1. Patients who refuse participation
2. Patients who are unable to receive or who refuse blood products
3. Patients who are involved in a preoperative autologous pre-donation program
4. Patients who are having a heart transplant or having surgery solely for an insertion of a ventricular assist device
5. Pregnancy or lactation (a negative pregnancy test must be obtained prior to randomization for women of childbearing potential)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Composite score of any one of the following events occurring 6 months after cardiac surgery: (1) all-cause mortality; (2) myocardial infarction; (3) new onset renal failure requiring dialysis; or (4) new focal neurological deficit (stroke). | Within 6 months after cardiac surgery.
  Any of all-cause mortality, myocardial infarction, new onset renal failure requiring dialysis, or new focal neurological deficit (stroke).

SECONDARY OUTCOMES:
Incidence of each individual component of the primary outcome: all-cause mortality, myocardial infarction, new onset renal failure requiring dialysis, and new focal neurological deficit (stroke). | Within 6 months after cardiac surgery.
  Incidence of all-cause mortality, myocardial infarction, new onset renal failure requiring dialysis, and new focal neurological deficit (stroke).
Composite and individual all-cause mortality, myocardial infarction, new onset renal failure requiring dialysis, and new focal neurological deficit (stroke). | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Composite and individual incidence of all-cause mortality, myocardial infarction, new onset renal failure requiring dialysis, and new focal neurological deficit (stroke).
Length of stay in the ICU and hospital. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Length of stay in the ICU and hospital in days.
Prolonged low output state. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Defined as the need for two or more inotropes for 24 hours or more, intra-aortic balloon pump or ventricular assist device postoperatively.
Duration of mechanical ventilation. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Time on mechanical ventilation.
Incidence of infection. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Defined as septic shock with positive blood cultures; pneumonia defined as autopsy diagnosis or roentgenographic infiltrate and at least two out of three of the following criteria: fever, leukocytosis, and positive sputum culture; and/or deep sternal or leg wound infection requiring intravenous antibiotics and/or surgical debridement.
Acute kidney injury. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Defined by the Kidney Disease Improving Global Outcomes (KDIGO) clinical practice guideline - a 50% increase in serum creatinine within 1 week or a 26.5 mmol/L increase within 48 hours.
Delirium. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Confusion Assessment Method (CAM) or CAM-ICU (even on 1 occasion), or Intensive Care Delirium Screening Checklist (ICDSC) > 3, or 3D-CAM, or 4AT ≥4, or more than one dose of haloperidol or similar antipsychotic drug, or documented delirium by neurologist or neurosurgeon or psychiatrist consultation.
Incidence of gut infarction. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Confirmed by imaging (e.g. angiography), autopsy, or through surgical means.
Hospital visits. | Within 6 months after cardiac surgery.
  Hospitalization and/or emergency visits and coronary revascularization after index procedure.
Transfusion requirements. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  The proportion of patients transfused and the number of blood products utilized (RBCs, plasma, platelets).
Incidence of seizures. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Generalized or focal tonic-clonic movements consistent with seizure; or electroencephalogram demonstrating epileptiform discharges; or diagnosis of seizures by neurologist or neurosurgeon consultation.
Incidence of encephalopathy. | Up to hospital discharge or after 28 days postoperatively, whichever comes first.
  Unexpected delayed awakening or severely altered mental status (unconscious despite no sedative medication for more than 5 days), or encephalopathy documented by neurologist or neurosurgeon or psychiatrist consultation.

CONTACTS AND LOCATIONS:
Overall Officials: David Mazer, MD, Principal Investigator — Unity Health Toronto; Nadine Shehata, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (54):
- United States (4):
  - Maine Medical Center, Portland, Maine
  - The Cooper Health System, Camden, New Jersey
  - Columbia University, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Australia (11):
  - Royal Adelaide Hospital, Adelaide, Adelaide
  - Royal Prince Alfred hospital, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne
  - Alfred Hospital, Prahran
- Canada (15):
  - University of Alberta Hospital, Edmonton, Alberta
  - Interior Health Kelowna General Hospital, Kelowna, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint John Regional Hospitall, Saint John, New Brunswick
  - Health Sciences North Research Institute, Greater Sudbury, Ontario
  - Hamilton Health Sciences Centre / Hamilton General Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hôpital Sacré-Cœur de Montréal, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumology de Québec - université Laval (IUCPQ-UL), Québec, Quebec
- Colombia (3):
  - Hospital Universitario San Ignacio, Bogotá
  - Fundacion Abood Shaio, Bogotá
  - Fundacion Cardioinfantil, Bogotá
- Nasr City Health Insurance Hospital, Naşr, Cairo Governorate, Egypt
- Democritus University of Thrace, Alexandroupoli, Evros, Greece
- EPIC Hospital, Ahmedabad, Gujarat, India
- Windhoek Central Hospital, Windhoek, Khomas Region, Namibia
- Shahid Gangalal National Heart Center, Kathmandu, Kathmandu, Nepal
- Emergency Institute of Cardiovascular Diseases, Bucharest, Romania, Romania
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia
- National Heart Centre, Singapore, Singapore
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa
- Spain (3):
  - Hospital de la Santa Creu I Sant Pau, Barcelona, Catalonia
  - Hospital General Universitari de Valencia, Valencia
  - Hospital Universitario La Fe Valencia, Valencia
- Switzerland (2):
  - Inselspital, University Hospital Bern, University of Bern, Bern, Canton of Bern
  - University Hospital Basel, Basel
- United Kingdom (7):
  - University Hospital Leicester, Leicester, East Midlands
  - Basildon University Hospitals-Mid and South Essex NHS Trust, Basildon, Essex
  - University Hospital Southampton Foundation Trust, Southampton, Hampshire
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Royal Papworth Hospital NHS Foundation Trust., Cambridge
  - Manchester University NHS Foundation Trust, Wythenshawe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836